CLINICAL TRIAL: NCT00143273
Title: Dose Response Study Of Lasofoxifene In Postmenopausal Women With Osteoporosis (Placebo-Controlled, Multicenter, Double-Blind, Comparative Study) - Japanese Asian Dose Evaluation: JADE
Brief Title: Dose Response Study of Lasofoxifene in Postmenopausal Women With Osteoporosis - Japanese Asian Dose Evaluation
Acronym: JADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Director, Project Management, Ligand Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A2181037
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Lasofoxifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Lasofoxifene Dose 1 (Experimental): 0.05 mg
  Interventions: Drug: lasofoxifene
- Lasofoxifene Dose 2 (Experimental): 0.25 mg
  Interventions: Drug: Lasofoxifene
- Lasofoxifene Dose 3 (Experimental): 0.5 mg
  Interventions: Drug: Lasofoxifene
- Placebo (Placebo Comparator): 0 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lasofoxifene — 0.05 mg tablets
  Arms: Lasofoxifene Dose 1
Drug: Placebo — 0 mg
  Arms: Placebo
Drug: Lasofoxifene — 0.25 mg tablets
  Arms: Lasofoxifene Dose 2
Drug: Lasofoxifene — 0.5 mg tablets
  Arms: Lasofoxifene Dose 3

SUMMARY:
To establish the optimal dose of lasofoxifene that is fully effective in increasing the BMD in postmenopausal Asian women.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal Asian women with osteoporosis defined by low BMD

Exclusion Criteria:

* Metabolic bone disease, use of other osteoporosis drugs or drugs interering with normal bone metabolism

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Effects of lasofoxifene compared to placebo on Bone Mineral Density (BMD) changes at the spine and hip after 1 year of treatment | 12 months
  Percent change from baseline in lumbar spine BMD at Month 12

SECONDARY OUTCOMES:
Hip BMD, bone markers, lipids and new radiographic vertebral fractures at 1 year | Month 6 and Month 12
  Percent change from baseline in lumbar spine BMD at Month 6, percent change in baseline in hip BMD at Month 6 and Month 12, percent change from baseline in bone metabolism markers at Month 6 and Month 12, percent change from baseline in serum lipids, total cholesterol, high-density lipoprotein cholesterol, triglycerides, lipoprotein (a), apoliporpotein-A1, apolipoprotein-B at Month 6 and Month 12 and incidence of new vertebral fractures at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Japan (8):
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kagoshima, Kagoshima-ken
  - Pfizer Investigational Site, Miyazaki, Miyazaki
  - Pfizer Investigational Site, Fuchū, Tokyo
  - Pfizer Investigational Site, Kiyose, Tokyo
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Yonago-shi, Tottori
- South Korea (3):
  - Pfizer Investigational Site, Kangnam-ku, Seoul
  - Pfizer Investigational Site, Sonpagu, Seoul
  - Pfizer Investigational Site, Youngdeungpo-gu, Seoul
- Taiwan (3):
  - Pfizer Investigational Site, Changhua
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyun 333
- Pfizer Investigational Site